CLINICAL TRIAL: NCT03545100
Title: Rehabilitation Outcomes of Shoulder Function in Oral Cancer Survivors Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201800026A3
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2019-08

CONDITIONS: Oral Cancer
Keywords: oral cancer; shoulder dysfunction; quality of life; motor control; strengthening exercise
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): motor control therapy
  Interventions: Other: motor control therapy; Other: regular physical therapy
- control group (Active Comparator): regular physical therapy
  Interventions: Other: regular physical therapy

INTERVENTIONS:
Other: motor control therapy — scapular muscle progressive resistive exercise(PRE)
  Arms: experimental group
Other: regular physical therapy — transcutaneous electrical nerve stimulation(TENS), shoulder joint ROM, scapular muscle PRE

SUMMARY:
Head and neck cancer is prevalent in Taiwan, and oral cancer is the most common location. Advanced treatment of oral cancer increases survival rates; however, it also increases the risk of developing shoulder dysfunction, dysphagia, oral dysfunction, donor site morbidity and psychological issues. The probability of shoulder dysfunction after neck dissection is as high as 70%. Rehabilitation effects on shoulder function for head and neck survivors are needed for further studied.The purpose of this randomized clinical trial is to explore the effects of rehabilitation for shoulder function in oral cancer survivors.

DETAILED DESCRIPTION:
Head and neck cancer is prevalent in Taiwan, and oral cancer is the most common location. Advanced treatment of oral cancer increases survival rates; however, it also increases the risk of developing shoulder dysfunction, dysphagia, oral dysfunction, donor site morbidity and psychological issues. The probability of shoulder dysfunction after neck dissection is as high as 70%. Rehabilitation effects on shoulder function for head and neck survivors are needed for further studied.

The purpose of this randomized clinical trial is to explore the effects of rehabilitation for shoulder function in oral cancer survivors. We will recruit 60 newly diagnosed oral cancer subjects through the plastic surgeon's referral from April 2018 to March 2020. The participants will be randomized separated into experimental or control group. Each group would receive regular physical therapy for shoulder function (i.e., transcutaneous electrical stimulation, shoulder joint range of motion exercise, scapular muscle strengthening training). Experimental group would be supplemented by motor control therapy targeting the scapular muscle progressive resistance exercise (exercise plus manual therapy).

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the inform consent
* Sufficiently communicate in the Chinese language
* Be able to follow instructions
* Newly diagnosed oral cancer
* Spinal accessory shoulder dysfunction

Exclusion Criteria:

* Pregnant or breast-feeding woman
* Cognitively impaired
* Central nervous disease
* Distant metastasis or recurrence
* A history of shoulder pain or known shoulder pathology
* Unable to communicate or comprehend the questionnaires

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
shoulder pain | 1 year
  Visual Analog Scale, the *total* range = 0-10
shoulder joint range of motion | 1 year
  abduction measured by goniometer
shoulder function | 1 year
  the Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure for upper extremity function
maximal isometric muscle strength | 1 year
  measurement for the upper trapezius, middle trapezius, lower trapezius and serrates anterior at the moment of SEMG

SECONDARY OUTCOMES:
surface electromyography (SEMG) | 1 year
  measure the muscle activities of the upper trapezius, middle trapezius, lower trapezius and serrates anterior
quality of life C-30 | 1 year
  European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30
quality of life H&N35 | 1 year
  European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-H&N35
return to work | 1 year
  duration between return-to-work and operation

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, Master, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Plastic and Reconstructive Surgery Rehabilitation Center, Chung Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Result] Wong CH, Wei FC. Microsurgical free flap in head and neck reconstruction. Head Neck. 2010 Sep;32(9):1236-45. doi: 10.1002/hed.21284. PMID 20014446
- [Result] Lutz BS, Wei FC. Microsurgical workhorse flaps in head and neck reconstruction. Clin Plast Surg. 2005 Jul;32(3):421-30, vii. doi: 10.1016/j.cps.2005.02.006. PMID 15979480
- [Result] Neligan PC. Head and neck reconstruction. Plast Reconstr Surg. 2013 Feb;131(2):260e-269e. doi: 10.1097/PRS.0b013e3182778938. PMID 23358022
- [Result] Pauloski BR, Rademaker AW, Logemann JA, Discekici-Harris M, Mittal BB. Comparison of swallowing function after intensity-modulated radiation therapy and conventional radiotherapy for head and neck cancer. Head Neck. 2015 Nov;37(11):1575-82. doi: 10.1002/hed.23796. Epub 2014 Aug 1. PMID 24909649
- [Result] Sheikh A, Shallwani H, Ghaffar S. Postoperative shoulder function after different types of neck dissection in head and neck cancer. Ear Nose Throat J. 2014 Apr-May;93(4-5):E21-6. PMID 24817237
- [Result] van der Molen L, van Rossum MA, Burkhead LM, Smeele LE, Rasch CR, Hilgers FJ. A randomized preventive rehabilitation trial in advanced head and neck cancer patients treated with chemoradiotherapy: feasibility, compliance, and short-term effects. Dysphagia. 2011 Jun;26(2):155-70. doi: 10.1007/s00455-010-9288-y. Epub 2010 Jul 11. PMID 20623305
- [Result] Eades M, Murphy J, Carney S, Amdouni S, Lemoignan J, Jelowicki M, Nadler M, Chasen M, Gagnon B. Effect of an interdisciplinary rehabilitation program on quality of life in patients with head and neck cancer: review of clinical experience. Head Neck. 2013 Mar;35(3):343-9. doi: 10.1002/hed.22972. Epub 2012 Mar 16. PMID 22422558
- [Result] McGarvey AC, Osmotherly PG, Hoffman GR, Chiarelli PE. Impact of neck dissection on scapular muscle function: a case-controlled electromyographic study. Arch Phys Med Rehabil. 2013 Jan;94(1):113-9. doi: 10.1016/j.apmr.2012.07.017. Epub 2012 Aug 1. PMID 22864015
- [Result] Hsieh LC, Chen JW, Wang LY, Tsang YM, Shueng PW, Liao LJ, Lo WC, Lin YC, Tseng CF, Kuo YS, Jhuang JY, Tien HJ, Juan HF, Hsieh CH. Predicting the severity and prognosis of trismus after intensity-modulated radiation therapy for oral cancer patients by magnetic resonance imaging. PLoS One. 2014 Mar 21;9(3):e92561. doi: 10.1371/journal.pone.0092561. eCollection 2014. PMID 24658376
- [Result] Wetzels JW, Merkx MA, de Haan AF, Koole R, Speksnijder CM. Maximum mouth opening and trismus in 143 patients treated for oral cancer: a 1-year prospective study. Head Neck. 2014 Dec;36(12):1754-62. doi: 10.1002/hed.23534. Epub 2014 Jan 30. PMID 24478217
- [Result] Lee R, Slevin N, Musgrove B, Swindell R, Molassiotis A. Prediction of post-treatment trismus in head and neck cancer patients. Br J Oral Maxillofac Surg. 2012 Jun;50(4):328-32. doi: 10.1016/j.bjoms.2011.06.009. Epub 2011 Jul 26. PMID 21794962
- [Result] Stubblefield MD. Radiation fibrosis syndrome: neuromuscular and musculoskeletal complications in cancer survivors. PM R. 2011 Nov;3(11):1041-54. doi: 10.1016/j.pmrj.2011.08.535. PMID 22108231
- [Result] Chan JY, Lua LL, Starmer HH, Sun DQ, Rosenblatt ES, Gourin CG. The relationship between depressive symptoms and initial quality of life and function in head and neck cancer. Laryngoscope. 2011 Jun;121(6):1212-8. doi: 10.1002/lary.21788. Epub 2011 May 3. PMID 21541945
- [Result] EWING MR, MARTIN H. Disability following radical neck dissection; an assessment based on the postoperative evaluation of 100 patients. Cancer. 1952 Sep;5(5):873-83. doi: 10.1002/1097-0142(195209)5:53.0.co;2-4. No abstract available. PMID 12988177
- [Result] Carr SD, Bowyer D, Cox G. Upper limb dysfunction following selective neck dissection: a retrospective questionnaire study. Head Neck. 2009 Jun;31(6):789-92. doi: 10.1002/hed.21018. PMID 19260131
- [Result] Dijkstra PU, van Wilgen PC, Buijs RP, Brendeke W, de Goede CJ, Kerst A, Koolstra M, Marinus J, Schoppink EM, Stuiver MM, van de Velde CF, Roodenburg JL. Incidence of shoulder pain after neck dissection: a clinical explorative study for risk factors. Head Neck. 2001 Nov;23(11):947-53. doi: 10.1002/hed.1137. PMID 11754498
- [Result] Erisen L, Basel B, Irdesel J, Zarifoglu M, Coskun H, Basut O, Tezel I, Hizalan I, Onart S. Shoulder function after accessory nerve-sparing neck dissections. Head Neck. 2004 Nov;26(11):967-71. doi: 10.1002/hed.20095. PMID 15459926
- [Result] Lima LP, Amar A, Lehn CN. Spinal accessory nerve neuropathy following neck dissection. Braz J Otorhinolaryngol. 2011 Mar-Apr;77(2):259-62. doi: 10.1590/s1808-86942011000200017. PMID 21537629
- [Result] Umeda M, Shigeta T, Takahashi H, Oguni A, Kataoka T, Minamikawa T, Shibuya Y, Komori T. Shoulder mobility after spinal accessory nerve-sparing modified radical neck dissection in oral cancer patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Jun;109(6):820-4. doi: 10.1016/j.tripleo.2009.11.027. Epub 2010 Mar 17. PMID 20299249
- [Result] Ishigaki T, Yamanaka M, Hirokawa M, Tai K, Ezawa Y, Samukawa M, Tohyama H, Sugawara M. Rehabilitation Exercises to Induce Balanced Scapular Muscle Activity in an Anti-gravity Posture. J Phys Ther Sci. 2014 Dec;26(12):1871-4. doi: 10.1589/jpts.26.1871. Epub 2014 Dec 25. PMID 25540485
- [Result] Cools AM, Dewitte V, Lanszweert F, Notebaert D, Roets A, Soetens B, Cagnie B, Witvrouw EE. Rehabilitation of scapular muscle balance: which exercises to prescribe? Am J Sports Med. 2007 Oct;35(10):1744-51. doi: 10.1177/0363546507303560. Epub 2007 Jul 2. PMID 17606671
- [Result] Andersen CH, Zebis MK, Saervoll C, Sundstrup E, Jakobsen MD, Sjogaard G, Andersen LL. Scapular muscle activity from selected strengthening exercises performed at low and high intensities. J Strength Cond Res. 2012 Sep;26(9):2408-16. doi: 10.1519/JSC.0b013e31823f8d24. PMID 22076101
- [Result] Cricchio M, Frazer C. Scapulothoracic and scapulohumeral exercises: a narrative review of electromyographic studies. J Hand Ther. 2011 Oct-Dec;24(4):322-33; quiz 334. doi: 10.1016/j.jht.2011.06.001. Epub 2011 Aug 5. PMID 21820276
- [Result] Worsley P, Warner M, Mottram S, Gadola S, Veeger HE, Hermens H, Morrissey D, Little P, Cooper C, Carr A, Stokes M. Motor control retraining exercises for shoulder impingement: effects on function, muscle activation, and biomechanics in young adults. J Shoulder Elbow Surg. 2013 Apr;22(4):e11-9. doi: 10.1016/j.jse.2012.06.010. Epub 2012 Sep 1. PMID 22947240
- [Result] McGarvey AC, Osmotherly PG, Hoffman GR, Chiarelli PE. Scapular muscle exercises following neck dissection surgery for head and neck cancer: a comparative electromyographic study. Phys Ther. 2013 Jun;93(6):786-97. doi: 10.2522/ptj.20120385. Epub 2013 Feb 21. PMID 23431215
- [Result] McNeely ML, Parliament MB, Seikaly H, Jha N, Magee DJ, Haykowsky MJ, Courneya KS. Effect of exercise on upper extremity pain and dysfunction in head and neck cancer survivors: a randomized controlled trial. Cancer. 2008 Jul 1;113(1):214-22. doi: 10.1002/cncr.23536. PMID 18457329
- [Result] Brown KE, Stickler L. Shoulder pain and dysfunction secondary to neural injury. Int J Sports Phys Ther. 2011 Sep;6(3):224-33. PMID 21904699
- [Result] McGarvey AC, Chiarelli PE, Osmotherly PG, Hoffman GR. Physiotherapy for accessory nerve shoulder dysfunction following neck dissection surgery: a literature review. Head Neck. 2011 Feb;33(2):274-80. doi: 10.1002/hed.21366. PMID 20222043
- [Result] Shepherd KL, Fisher SE. Prospective evaluation of quality of life in patients with oral and oropharyngeal cancer: from diagnosis to three months post-treatment. Oral Oncol. 2004 Aug;40(7):751-7. doi: 10.1016/j.oraloncology.2004.01.018. PMID 15172646
- [Result] Schliephake H, Jamil MU. Prospective evaluation of quality of life after oncologic surgery for oral cancer. Int J Oral Maxillofac Surg. 2002 Aug;31(4):427-33. doi: 10.1054/ijom.2001.0194. PMID 12361079
- [Result] Barrios R, Bravo M, Gil-Montoya JA, Martinez-Lara I, Garcia-Medina B, Tsakos G. Oral and general health-related quality of life in patients treated for oral cancer compared to control group. Health Qual Life Outcomes. 2015 Jan 23;13:9. doi: 10.1186/s12955-014-0201-5. PMID 25613348
- [Result] McNeely ML, Parliament MB, Seikaly H, Jha N, Magee DJ, Haykowsky MJ, Courneya KS. Sustainability of outcomes after a randomized crossover trial of resistance exercise for shoulder dysfunction in survivors of head and neck cancer. Physiother Can. 2015 Winter;67(1):85-93. doi: 10.3138/ptc.2014-13O. PMID 25931658
- [Result] Ch'ng S, Oates J, Gao K, Foo K, Davies S, Brunner M, Clark JR. Prospective quality of life assessment between treatment groups for oral cavity squamous cell carcinoma. Head Neck. 2014 Jun;36(6):834-40. doi: 10.1002/hed.23387. Epub 2013 Sep 2. PMID 23720248
- [Result] McGarvey AC, Hoffman GR, Osmotherly PG, Chiarelli PE. Maximizing shoulder function after accessory nerve injury and neck dissection surgery: A multicenter randomized controlled trial. Head Neck. 2015 Jul;37(7):1022-31. doi: 10.1002/hed.23712. Epub 2014 Jul 11. PMID 25042422
- [Result] Chan JY, Wong ST, Chan RC, Wei WI. Shoulder Dysfunction after Selective Neck Dissection in Recurrent Nasopharyngeal Carcinoma. Otolaryngol Head Neck Surg. 2015 Sep;153(3):379-84. doi: 10.1177/0194599815590589. Epub 2015 Jul 2. PMID 26138607
- [Result] Cranney A, Welch V, Wells G, Adachi J, Shea B, Simon L, Tugwell P. Discrimination of changes in osteoporosis outcomes. J Rheumatol. 2001 Feb;28(2):413-21. PMID 11246689
- [Result] Beaton DE, Bombardier C, Katz JN, Wright JG, Wells G, Boers M, Strand V, Shea B. Looking for important change/differences in studies of responsiveness. OMERACT MCID Working Group. Outcome Measures in Rheumatology. Minimal Clinically Important Difference. J Rheumatol. 2001 Feb;28(2):400-5. PMID 11246687
- [Result] Canis M, Weiss BG, Ihler F, Hummers-Pradier E, Matthias C, Wolff HA. Quality of life in patients after resection of pT3 lateral tongue carcinoma: Microvascular reconstruction versus primary closure. Head Neck. 2016 Jan;38(1):89-94. doi: 10.1002/hed.23862. Epub 2015 Jun 16. PMID 25224592
- [Result] Bjordal K, Hammerlid E, Ahlner-Elmqvist M, de Graeff A, Boysen M, Evensen JF, Biorklund A, de Leeuw JR, Fayers PM, Jannert M, Westin T, Kaasa S. Quality of life in head and neck cancer patients: validation of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-H&N35. J Clin Oncol. 1999 Mar;17(3):1008-19. doi: 10.1200/JCO.1999.17.3.1008. PMID 10071296
- [Result] Chie WC, Hong RL, Lai CC, Ting LL, Hsu MM. Quality of life in patients of nasopharyngeal carcinoma: validation of the Taiwan Chinese version of the EORTC QLQ-C30 and the EORTC QLQ-H&N35. Qual Life Res. 2003 Feb;12(1):93-8. doi: 10.1023/a:1022070220328. PMID 12625522
- [Result] Sherman AC, Simonton S, Adams DC, Vural E, Owens B, Hanna E. Assessing quality of life in patients with head and neck cancer: cross-validation of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Head and Neck module (QLQ-H&N35). Arch Otolaryngol Head Neck Surg. 2000 Apr;126(4):459-67. doi: 10.1001/archotol.126.4.459. PMID 10772298
- [Derived] Chen YH, Huang CY, Liang WA, Lin CR, Chao YH. Effects of Conscious Control of Scapular Orientation in Oral Cancer Survivors With Scapular Dyskinesis: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211040827. doi: 10.1177/15347354211040827. PMID 34412536